CLINICAL TRIAL: NCT03533153
Title: Clinical Study on Ischemia-Reperfusion Injury Using Intravenous Administration of MSC in Patients With Myocardial Infarction Intended to Improve MVO and Prognosis After Surgery
Brief Title: Intravenous MSC Therapy on Ischemia-Reperfusion Injury in Patients With Myocardial Infarction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Biao Xu, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSC-NanjingUMS
Record Dates: First submitted 2018-01-24; First posted 2018-05-23 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Myocardial Infarction
Keywords: MSC
MeSH Terms: conditions — Myocardial Infarction | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WJ-MSC cells implantation group (Experimental): MSC cells (allogeneic transplantation from WJ-MSC primary cells); the frequency: for one time within12h after emergency coronary artery revascularization; dose levels: 1X10^8; method of administration: intravenous injection. Other kinds of treatment are in accordance with the treatment guidelines for MI patients, listed in the column "Conventional drug therapy".
  Interventions: Biological: WJ-MSC cells implantation; Drug: Conventional drug therapy
- CTSTMD PBS without WJ-MSC group (Placebo Comparator): Saline only was injected in the control group. The frequency: for one time 2-12h after emergency coronary artery revascularization. Dose levels: the same dosage given to MSC group. Method of administration: intravenous injection. Other kinds of treatment are in accordance with the treatment guidelines for MI patients, listed in the column "Conventional drug therapy".
  Interventions: Drug: CTSTMD PBS without WJ-MSC; Drug: Conventional drug therapy

INTERVENTIONS:
Biological: WJ-MSC cells implantation — Laboratory of Stem Cell of Drum Tower Hospital, Nanjing University Medical School, is able to provide types of Good Manufacture Practice (GMP) level stem cells and stem cell-based medicinal products. Clinical-grade WJ-MSC primary cells are cultured to 4~ 8 passages, and the surface markers (CD90+, CD105+, CD45-, CD31-, CD117-) are identified by flow cytometry. WJ-MSC cells are trypsinized and resuspended in the wash buffer of CTSTMD PBS (+Ca2+, +Mg2+). Within 2 hours after enzyme digestion, WJ-MSC cells are shipped to coronary care unit (CCU) and injected into the body.
  Other Names: WJ-MSC
  Arms: WJ-MSC cells implantation group
Drug: CTSTMD PBS without WJ-MSC — For Case-control study only.
  Other Names: CTSTMD PBS
  Arms: CTSTMD PBS without WJ-MSC group
Drug: Conventional drug therapy — All patients undergo guideline-recommended treatment for STEMI, including aspirin (loading dose of 300mg before maintenance dose of 100 mg/d), clopidogrel (loading dose of 300mg before maintenance dose of 75 mg/d) or Ticagrelor (loading dose of 300mg before maintenance dose of 90 mg/d), angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB), β-receptor blockers, statins and nitrate esters.
  Other Names: Conventional

SUMMARY:
The investigators scheduled to assess the value of intravenous injection of WJ-MSC in patients with ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
Ischemia/reperfusion injury in myocardial infarction can induce mass release of oxygen free radicals, trigger inflammatory reaction, and ultimately lead to myocardial remodeling and irreversible cardiac function decline. Microvascular obstruction (MVO) and haemorrhage are common pathological alternations in myocardium post primary PCI, which provide strong prognostic information for STEMI patients. Till now, there is no treatment to be used in clinical practice to reduce myocardium MVO and haemorrhage. With the deep research on stem cells, it is found that the benefits of MSC transplants for myocardium infarction may be achieved by its paracrine effect. Meanwhile, the immunoregulatory effect of MSC has been widely reported in multiply immune disease. Therefore, the applicant proposed the hypothesis that MSC can play an effective role in reducing oxidative stress and inflammatory response, inhibiting microvascular obstruction and haemorrhage. Intravenous injection of MSC will be used in patients with STEMI within 12 hours post primary PCI. The primary endpoint and safety endpoint are recorded in the one year follow up to assess the clinical outcome of intravenous MSC treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75;
2. First performance of anterior acute ST-segment elevation myocardial infarction (STEMI), Killip grade 2 or below on admission;
3. Completing emergency percutaneous coronary intervention within 12h, with TIMI flow grade 0 or 1 (before stent implantation) and 3 (after stent implantation);
4. LVEF in echocardiography is 45% or below primary PCI.

Exclusion Criteria:

1. Medical history of Q wave myocardial infarction, significant valve disease, pericarditis, pericardial tamponade, myocardiopathy, chronic heart failure or cardio embolism;
2. Non ST-segment elevation myocardial infarction;
3. Chronic occlusion in LCX or RCA besides LAD;
4. Diagnosed with severe coronary artery disease but not yet causing a loss of heart function;
5. Hemodynamic disorders, shock or respiratory failure on admission;
6. Atrial fibrillation with warfarin treatment only or at high risk of bleeding;
7. Constant tachycardia, malignant arrhythmia, complete atrioventricular block, new-onset complete left bundle branch block (LBBB) or pacemaker implantation;
8. Mechanical complications of acute myocardial infarction (interventricular septal defect, rupture of papillary muscle, etc.) or huge left ventricular aneurysm could only be corrected through surgical procedures;
9. Chronic pulmonary heart disease (COPD, bronchial asthma, chronic bronchitis, emphysema or pulmonary heart disease), autoimmune disease or patients on immunosuppressive therapy;
10. Acute infective disease;
11. Hepatitis B/C virus or HIV;
12. Blood system diseases (thrombocytopenia, severe anemia, leukemia, etc.);
13. Severe renal insufficiency, with creatinine clearance (CCr) <33 ml/min or serum creatinine >133 μmol/L;
14. Obvious abnormalities in liver function (ALT and AST 3 times higher than the upper limit of normal value);
15. Medical history of cerebral hemorrhage;
16. Medical history of the malignant tumor;
17. Cognitive impairment, dementia or severe mental illness (SMI);
18. Substantial disability negatively influenced regular follow-up research;
19. Systematic diseases not been effectively controlled or life expectancy < 1 year;
20. Pregnant or lactating women;
21. Not suitable for MRI examination, or could not stick to treatment plans;
22. Could not or not willing to give written informed consent.

Exit Criteria:

1. Intolerable infaust events or changed treatment strategy leading to serious violations of trial conduct;
2. Requiring to exit the clinical trial;
3. Research scheme violations, severely disrupted safety and effectiveness of the trail;
4. Lost to follow-up cases;
5. Conceiving children or want to do that during the treatment period;
6. Candidates not fit to carry on the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
IS | at Month 3 after treatment.
  The primary endpoint is based on patients' myocardial infarction size (IS) as a result of CMR examination. The detection is recorded in the follow up at Month 3.

SECONDARY OUTCOMES:
MACCE | within 1 year after PCI.
  Follow up main adverse cardiovascular and cerebrovascular events (MACCE) such as death, myocardial infarction, stroke and heart failure within 1 year after treatment.
MVO and Hemorrhage | at Day 4 to Day 7 after PCI.
  Patients underwent cardiac magnetic resonance imaging (CMR) at Day 4 to Day 7 after presentation with STEMI on a 3.0-T scanner.The change in Microvascular obstruction (MVO) and intramyocardial hemorrhage would be followed up. MVO was defined (and quantified) as hypoenhancement within infarcted myocardium, as determined from LGE images, and was included in the total infarct size. Myocardial oedema was quantified using semi-automatic thresholding, defining AAR as enhancement within myocardium of signal intensity > 2 standard deviations (SDs) above that of a region of interest contoured in remote myocardium. Hypoenhanced areas within the AAR were regarded as intramyocardial haemorrhage (IMH). The MSI was calculated as 100 × [(AAR - infarct size)/AAR]. Infarct size, MVO, AAR and IMH were expressed as %LVM and LV volumes were indexed to body surface area.
CMR Markers of Myocardial and Microvascular Damage | at Month 3 after PCI.
  CMR markers of myocardial and microvascular damage (myocardial salvage, left ventricular end diastolic volume (LVEDV), left ventricular ejection fraction (LVEF), microvascular obstruction (MVO), intramyocardial hemorrhage) would be followed up at Month 3 after treatment.
CK-MB and Troponin | at baseline and at Hour 6, Hour 12, Hour 24 and Hour 48 after PCI.
  A sensitive troponin T assay for the early diagnosis and risk stratification of myocardial infarction would be evaluated. Blood samples were drawn at baseline and at Hour 6, Hour 12, Hour 24 and Hour 48 after PPCI for cardiac enzyme [creatine kinase MB isoenzyme (CK-MB) and troponin] estimation
Echocardiographic Changes | at Hour 6, Week 1, Month 1, Month 6 and Year 1 after PCI.
  Changes in echocardiography would be tested at Hour 6, Week 1, Month 1, Month 6 and Year 1 after treatment.
6-min Walk Test | at Hour 6, Week1, Month 1, Month 6 and Year 1 after PCI.
  Changes in 6-min walk test would be tested at Hour 6, Week1, Month 1, Month 6 and Year 1 after treatment.
Serum BNP | at Hour 7, Month 1, Month 6 and Year 1 after PCI.
  Changes in patients' serum BNP level would be tested at Hour 7, Month 1, Month 6 and Year 1 after treatment.
MLHFQ Scale | at Week1, Month 1, Month 6 and Year 1 after PCI.
  Patients would be required to fill out the quality of life (QQL) scale Minnesota Living with Heart Failure Questionnaire (MLHFQ) at Week1, Month 1, Month 6 and Year 1 after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: BIAO XU, Ph.D., Study Chair — Drum Tower Hospital, Nanjing University Medical School

IPD SHARING:
Plan to Share IPD: No
We have not decided to make it open.

REFERENCES:
- [Background] Ahn JM, Park DW, Lee CW, Chang M, Cavalcante R, Sotomi Y, Onuma Y, Tenekecioglu E, Han M, Lee PH, Kang SJ, Lee SW, Kim YH, Park SW, Serruys PW, Park SJ. Comparison of Stenting Versus Bypass Surgery According to the Completeness of Revascularization in Severe Coronary Artery Disease: Patient-Level Pooled Analysis of the SYNTAX, PRECOMBAT, and BEST Trials. JACC Cardiovasc Interv. 2017 Jul 24;10(14):1415-1424. doi: 10.1016/j.jcin.2017.04.037. PMID 28728654
- [Background] Symons R, Pontone G, Schwitter J, Francone M, Iglesias JF, Barison A, Zalewski J, de Luca L, Degrauwe S, Claus P, Guglielmo M, Nessler J, Carbone I, Ferro G, Durak M, Magistrelli P, Lo Presti A, Aquaro GD, Eeckhout E, Roguelov C, Andreini D, Vogt P, Guaricci AI, Mushtaq S, Lorenzoni V, Muller O, Desmet W, Agati L, Janssens S, Bogaert J, Masci PG. Long-Term Incremental Prognostic Value of Cardiovascular Magnetic Resonance After ST-Segment Elevation Myocardial Infarction: A Study of the Collaborative Registry on CMR in STEMI. JACC Cardiovasc Imaging. 2018 Jun;11(6):813-825. doi: 10.1016/j.jcmg.2017.05.023. Epub 2017 Aug 16. PMID 28823746
- [Background] Cuculi F, Dall'Armellina E, Manlhiot C, De Caterina AR, Colyer S, Ferreira V, Morovat A, Prendergast BD, Forfar JC, Alp NJ, Choudhury RP, Neubauer S, Channon KM, Banning AP, Kharbanda RK. Early change in invasive measures of microvascular function can predict myocardial recovery following PCI for ST-elevation myocardial infarction. Eur Heart J. 2014 Aug 1;35(29):1971-80. doi: 10.1093/eurheartj/eht434. Epub 2013 Oct 17. PMID 24135835
- [Background] Robbers LF, Eerenberg ES, Teunissen PF, Jansen MF, Hollander MR, Horrevoets AJ, Knaapen P, Nijveldt R, Heymans MW, Levi MM, van Rossum AC, Niessen HW, Marcu CB, Beek AM, van Royen N. Magnetic resonance imaging-defined areas of microvascular obstruction after acute myocardial infarction represent microvascular destruction and haemorrhage. Eur Heart J. 2013 Aug;34(30):2346-53. doi: 10.1093/eurheartj/eht100. Epub 2013 Apr 17. PMID 23594591